CLINICAL TRIAL: NCT01896869
Title: A Phase 2, Multicenter Study of FOLFIRINOX Followed by Ipilimumab in Combination With Allogeneic GM-CSF Transfected Pancreatic Tumor Vaccine in the Treatment of Metastatic Pancreatic Cancer
Brief Title: FOLFIRINOX Followed by Ipilimumab With Pancreatic Tumor Vaccine in Treatment of Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J13108; NA_00086350 (Other: JHMIRB); FD-R-004819-01 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2020-05-06 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: Pancreatic Cancer; Vaccine; Immunotherapy; Ipilimumab; cytotoxic T-lymphocyte-associated protein 4 (CTLA-4); antibody; FOLFIRINOX
MeSH Terms: conditions — Pancreatic Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Ipilimumab; Vaccines; folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab + Vaccine (Arm A) (Experimental): Ipilimumab and vaccine will be administered every 3 weeks for 4 doses, then every 8 weeks.
  Interventions: Drug: Ipilimumab; Biological: Vaccine
- FOLFIRINOX (Arm B) (Experimental): Administered every 14 days (one cycle)
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: Ipilimumab — 3 mg/kg administered IV (10mg/kg if treatment started prior to protocol v 6.3)
  Other Names: MDX-010; BMS-734016
  Arms: Ipilimumab + Vaccine (Arm A)
Biological: Vaccine — 5x10^8 cells administered in 6 intradermal injections
  Other Names: PANC 6.03 pcDNA-1/GM-Neo and PANC 10.05 pcDNA-1/GM-Neo; Allogeneic GM-CSF-Transduced Pancreatic Tumor Cell Vaccine (GVAX)
  Arms: Ipilimumab + Vaccine (Arm A)
Drug: FOLFIRINOX — Standard of care FOLFIRINOX may be modified according to the patient's known tolerability. Acceptable modified options could include 5-FU alone, capecitabine, FOLFOX, FOLFIRI, or FOLFIRINOX on a 21 day cycle.
  Arms: FOLFIRINOX (Arm B)

SUMMARY:
This study will enroll patients who have metastatic pancreatic cancer with stable disease on FOLFIRINOX chemotherapy. The main purpose of this study is to compare survival between patients that receive ipilimumab and a pancreatic tumor vaccine and patients who continue to receive FOLFIRINOX.

Funding Source - FDA Office of Orphan Product Development (OOPD)

ELIGIBILITY:
Inclusion Criteria (abbreviated):

1. Documented adenocarcinoma of the pancreas
2. Stable metastatic pancreatic cancer after 8-12 doses of FOLFIRINOX
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Life expectancy greater than 3 months
5. Adequate organ and marrow function defined by study-specified laboratory tests.
6. Must use acceptable form of birth control while on study
7. Oxygen saturation on room air >92%

Exclusion Criteria (abbreviated):

1. Surgery within 4 weeks of dosing investigational agent (some exceptions for minor procedures)
2. Off FOLFIRINOX treatment for more than 70 days prior to treatment on study
3. Prior chemotherapy for metastatic pancreatic cancer (other than FOLFIRINOX or adjuvant therapy).
4. History of prior treatment with ipilimumab, anti-PD1 antibody, CD137 agonist, or anti-CD40 antibody
5. Received any non-oncology live vaccine therapy up to one month prior to or after any dose of ipilimumab/vaccine
6. Receiving any other investigational agents
7. Any of the following concomitant therapy: IL-2, interferon, immunosuppressive agents, or chronic use of systemic corticosteroids
8. History of symptomatic autoimmune disease or immune impairment. Thyroid disease is allowed.
9. Known brain metastasis
10. Radiographic ascites that is apparent on physical exam or requiring intervention in the 2 months prior to enrollment
11. Uncontrolled intercurrent illness
12. Known or suspected hypersensitivity to GM-CSF
13. Chronic HIV, Hepatitis B or Hepatitis C
14. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dung Le, M.D., Principal Investigator — The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ipilimumab + Vaccine: Ipilimumab and vaccine will be administered every 3 weeks for 4 doses, then every 8 weeks.
  Ipilimumab: 3 mg/kg administered IV (10mg/kg if treatment started prior to protocol v 6.3)
  Vaccine: 5x10^8 cells administered in 6 intradermal injections
- FOLFIRINOX: Administered every 14 days (one cycle)
  FOLFIRINOX: Standard of care FOLFIRINOX may be modified according to the patient's known tolerability. Acceptable modified options could include 5-FU alone, capecitabine, FOLFOX, FOLFIRI, or FOLFIRINOX on a 21 day cycle.
Period: Overall Study
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Started | 41 | 42
Completed | 40 | 36
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 0 | 6
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX | Total
Number analyzed (Participants) | 41 | 42 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 26 | 56
  >=65 years | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 24 | 26 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 41 | 39 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 36 | 36 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
CA19-9 Secretors [Count of Participants; unit: Participants] — Carbohydrate Antigen 19-9 (CA19-9) is a tumor marker measured in the blood of patients with pancreas cancer. Not all patients with pancreas cancer will have elevated CA19-9 and there are some conditions other than cancer that can cause an elevated CA19-9. Normal CA19-9 range is 0- 36 U/mL. Individuals with elevated CA19-9 were considered secretors. Those who did not express CA19-9 were considered non-secretors.
  Participants | 32 | 31 | 63
CA19-9 at baseline [Median (Inter-Quartile Range); unit: IU/mL] — Carbohydrate Antigen 19-9 (CA19-9) is a tumor marker measured in the blood of patients with pancreas cancer. Not all patients with pancreas cancer will have elevated CA19-9 and there are some conditions other than cancer that can cause an elevated CA19-9. Normal CA19-9 range is 0- 36 U/mL. Population: Individuals who did not express CA19-9 were considered non-secretors and were excluded from analysis.
  IU/mL
    number analyzed (Participants) | 32 | 31 | 63
    (all) | 185.0 [46.0 to 1091.5] | 85.0 [41.6 to 178.7] | 117.1 [44.7 to 372.6]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall Survival is the time between the date of randomization on study and death.
Time Frame: 4 years
Population: 1 Arm A (Ipilimumab + Vaccine) patient was lost to follow-up prior to treatment and was excluded from analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 40 | 42
Months | 9.38 [5.0 to 12.2] | 14.7 [11.6 to 20.0]

2. Secondary Outcome: Toxicity of Ipilimumab in Combination With Pancreatic Tumor Vaccine
Description: Toxicity was assessed as the number of patients experiencing study drug-related adverse events (AEs). Data reported for only study drug-related adverse events (not all adverse events as reported in the adverse events section).
Time Frame: From the first dose of study drug through 70 days after last dose, up to 13 months
Population: AEs were not collected for Arm B subjects (FOLFIRINOX). 39 Arm A subjects (Ipilimumab+Vaccine) received at least 1 dose of study drug and were evaluable for toxicity. Dose of Ipilimumab was reduced from 10 mg/kg to 3 mg/kg due to toxicity concerns. Toxicity rates are compared between these dosing subgroups.
Measure: Count of Participants; unit: Participants
Groups:
- 3 mg/kg: Ipilimumab and vaccine administered every 3 weeks for 4 doses, then every 8 weeks.
  Ipilimumab: 3 mg/kg administered IV
  Vaccine: 5x10^8 cells administered in 6 intradermal injections
- 10 mg/kg: Ipilimumab and vaccine administered every 3 weeks for 4 doses, then every 8 weeks.
  Ipilimumab: 10 mg/kg administered IV
  Vaccine: 5x10^8 cells administered in 6 intradermal injections
Arm/Group | 3 mg/kg | 10 mg/kg
Number analyzed (Participants) | 14 | 25
Participants
  Any study drug-related AE | 13 | 25
  adrenal insufficiency | 0 | 1
  alopecia | 0 | 1
  ALT increased | 0 | 2
  arthralgia | 0 | 2
  AST increased | 0 | 1
  chills | 2 | 5
  colitis | 1 | 4
  cough | 0 | 1
  diarrhea | 1 | 2
  dry mouth | 0 | 1
  dry skin | 1 | 0
  edema face | 0 | 1
  fatigue | 1 | 7
  fever | 3 | 11
  flu-like symptoms | 1 | 2
  flushing | 0 | 1
  hepatitis | 0 | 1
  hyperhidrosis | 0 | 2
  hypophysitis | 1 | 2
  hypotension | 0 | 1
  hypothyroidism | 0 | 1
  lymph node pain | 0 | 2
  lymph node swelling | 0 | 1
  malaise | 1 | 0
  myalgia | 2 | 0
  nausea | 1 | 2
  pneumonitis | 0 | 1
  pruritus | 2 | 7
  rash | 8 | 18
  swelling, chest wall mass | 0 | 1
  thyroiditis | 0 | 1
  urticaria | 2 | 1
  vomiting | 1 | 2
  weight loss | 0 | 1
  vaccine site blisters | 1 | 4
  vaccine site bruising | 1 | 2
  vaccine site erythema | 11 | 20
  vaccine site flares | 0 | 2
  vaccine site induration | 12 | 25
  vaccine site oozing | 0 | 1
  vaccine site pruritus | 11 | 22
  vaccine site scabbing | 0 | 1
  vaccine site tenderness | 3 | 13

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is the time from date of randomization to progression or death, whichever comes first. Individuals without follow-up scans were censored one day after randomization and individuals with follow-up scans who did not have disease progression were censored at date of last scan.
Time Frame: Up to 4 years
Population: 1 Arm A patient was lost to follow-up prior to treatment and was excluded from analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 40 | 42
Months | 2.40 [1.87 to 2.53] | 5.55 [3.32 to 8.51]

4. Secondary Outcome: Immune-related Progression Free Survival (irPFS)
Description: Immune-related Progression Free Survival is the median time from date of randomization to disease progression or death, whichever comes first. Individuals without follow-up scans were censored one day after randomization and individuals with follow-up scans who did not have disease progression were censored at date of last scan.
  Disease progression was evaluated using immune-related Response Criteria (irRC). irRC differs from RECIST primarily in that target lesions are measured in 2 dimensions and new lesions contribute to tumor burden, but do not by themselves qualify as progressive disease.
Time Frame: Up to 4 years
Population: 1 Arm A patient was lost to follow-up prior to treatment and was excluded from analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 40 | 42
Months | 2.50 [2.14 to 2.92] | 5.55 [3.38 to 8.51]

5. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the number of patients from each group achieving a Complete Response (CR) or Partial Response (PR) by Response Evaluation Criteria In Solid Tumors (RECIST).
Time Frame: Assessed until disease progression, up to 2 years
Population: 6 Arm A patients were excluded from analysis (1 lost to follow-up prior to treatment, 1 off study before first follow-up scan, 4 had no measurable disease at baseline and therefore could not have a radiographic response). 13 Arm B patients were excluded from analysis (7 came off study before first follow-up scan, 6 had no measurable disease)
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 35 | 29
Participants | 1 | 3

6. Secondary Outcome: Immune-related Objective Response Rate
Description: Immune-related Objective Response Rate (irORR) is measured the same way, except that tumor responses are evaluated using immune-related response criteria (irRC).
  irRC differs from RECIST primarily in that target lesions are measured in 2 dimensions and new lesions contribute to tumor burden, but do not by themselves qualify as progressive disease.
Time Frame: Assessed until disease progression, up to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 35 | 29
Participants | 2 | 4

7. Secondary Outcome: Duration of Response
Description: Average length of time between achieving a complete response (CR) or partial response (PR) and documentation of recurrent or progressive disease.
Time Frame: Up to 22 months
Population: Only 1 patient on Arm A (Ipilimumab + Vaccine) and 3 patients on Arm B (FOLFIRINOX) achieved a response by RECIST and were included in this analysis. 2 additional patients (1 Arm A and 1 Arm B) achieved a response by irRC, but these patients were both taken off study the same day as their partial response, for disease progression by RECIST.
Measure: Mean (Full Range); unit: months
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 1 | 3
months | 2.5 [2.5 to 2.5] | 8.49 [2.73 to 17.45]

8. Secondary Outcome: Tumor Marker Kinetics as Assessed by Median Carbohydrate Antigen 19-9 (CA19-9) Levels
Description: Carbohydrate Antigen 19-9 (CA19-9) is a tumor marker measured in the blood of patients with pancreas cancer. Not all patients with pancreas cancer will have elevated CA19-9 and there are some conditions other than cancer that can cause an elevated CA19-9. Normal CA19-9 range is 0-36 U/mL.
Time Frame: Baseline, Week 7, and Week 10 visits
Population: Only patients who were considered CA19-9 secretors (expressed CA19-9 either on study or prior to study) were included in the analysis. 32 in Arm A (Ipilimumab+Vaccine) and 31 in Arm B (FOLFIRINOX). Only subjects evaluable for this outcome at the specified time points had CA19-9 drawn and could be included in the analysis.
Measure: Median (Inter-Quartile Range); unit: IU/mL
Groups:
- Ipilimumab + Vaccine: Ipilimumab and vaccine administered every 3 weeks for 4 doses, then every 8 weeks.
  Ipilimumab: 3 mg/kg administered IV (10mg/kg if treatment started prior to protocol v 6.3)
  Vaccine: 5x10^8 cells administered in 6 intradermal injections
Arm/Group | Ipilimumab + Vaccine | FOLFIRINOX
Number analyzed (Participants) | 32 | 31
IU/mL
  Baseline | 185.0 [46.0 to 1091.5] | 85.0 [41.6 to 178.7]
  Week 7: number analyzed (Participants) | 26 | 21
  Week 7 | 189.2 [61.2 to 7123.7] | 77.9 [23.4 to 430.0]
  Week 10: number analyzed (Participants) | 18 | 15
  Week 10 | 237.1 [64.4 to 4690.1] | 66.8 [24.0 to 443.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the first dose of study drug through 70 days after the last dose of study drug, up to 13 months
Description: AEs were not collected for Arm B subjects (FOLFIRINOX). 39 Arm A subjects (Ipilimumab+Vaccine) received at least 1 dose of study drug and were evaluable for toxicity.
Arm/Group | Ipilimumab + Vaccine
All-Cause Mortality (participants affected / at risk) | 5/39
Serious Adverse Events (participants affected / at risk) | 20/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Vaccine (N=39)
abdominal pain (Gastrointestinal disorders) | 2
acute kidney injury (Renal and urinary disorders) | 1
adrenal insufficiency (Endocrine disorders) | 1
alkaline phosphatase increased (Investigations) | 1
bacteremia (Infections and infestations) | 1
blood bilirubin increased (Investigations) | 2
catheter related infection (Infections and infestations) | 1
chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1
colitis (Gastrointestinal disorders) | 3
death, disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
delerium (Psychiatric disorders) | 1
diarrhea (Gastrointestinal disorders) | 2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
hypophysitis (Endocrine disorders) | 1
INR increased (Investigations) | 1
lung infection (Infections and infestations) | 2
malabsorption (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 1
neutropenia (Investigations) | 1
obstruction gastric (Gastrointestinal disorders) | 1
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
sepsis (Infections and infestations) | 2
platelet count decreased (Investigations) | 1
thromboembolic event - pulmonary embolism (Vascular disorders) | 1
vomiting (Gastrointestinal disorders) | 2
weight loss (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + Vaccine (N=39)
abdominal distention (Gastrointestinal disorders) | 3
abdominal pain (Gastrointestinal disorders) | 13
alkaline phosphatase increased (Investigations) | 3
alanine aminotransferase (ALT) increased (Investigations) | 5
anemia (Investigations) | 4
anorexia (Metabolism and nutrition disorders) | 9
anxiety (Psychiatric disorders) | 7
arthralgia (Musculoskeletal and connective tissue disorders) | 6
ascites (Gastrointestinal disorders) | 5
aspartate aminotransferase (AST) increased (Investigations) | 3
atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
back pain (Musculoskeletal and connective tissue disorders) | 7
bloating (Gastrointestinal disorders) | 5
blood bilirubin increased (Investigations) | 2
bruising (Injury, poisoning and procedural complications) | 4
chills (General disorders) | 12
cold intolerance (General disorders) | 2
colitis (Gastrointestinal disorders) | 4
constipation (Gastrointestinal disorders) | 14
cough (Respiratory, thoracic and mediastinal disorders) | 6
depression (Psychiatric disorders) | 3
diarrhea (Gastrointestinal disorders) | 12
difficulty urinating (Renal and urinary disorders) | 2
dizziness (Nervous system disorders) | 4
dry mouth (Gastrointestinal disorders) | 3
dry skin (Skin and subcutaneous tissue disorders) | 2
dyspepsia (Gastrointestinal disorders) | 3
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
edema limbs (General disorders) | 5
fall (Injury, poisoning and procedural complications) | 2
fatigue (General disorders) | 17
fever (General disorders) | 20
flatulence (Gastrointestinal disorders) | 2
flu-like symptoms (General disorders) | 3
gait disturbance (General disorders) | 2
headache (Nervous system disorders) | 6
hot flashes (Vascular disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 2
hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
hypokalemia (Metabolism and nutrition disorders) | 2
hypophosphatemia (Metabolism and nutrition disorders) | 2
hypophysitis (Endocrine disorders) | 3
hypotension (Vascular disorders) | 5
insomnia (Psychiatric disorders) | 12
lymph node pain (Blood and lymphatic system disorders) | 2
lymphocyte count decreased (Investigations) | 2
muscle cramp (Musculoskeletal and connective tissue disorders) | 3
myalgia (Musculoskeletal and connective tissue disorders) | 2
nausea (Gastrointestinal disorders) | 12
non-cardiac pain (General disorders) | 5
oral pain (Gastrointestinal disorders) | 2
pain, site of procedure/conmed (Injury, poisoning and procedural complications) | 3
peripheral sensory neuropathy (Nervous system disorders) | 2
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
pruritus (Skin and subcutaneous tissue disorders) | 9
rash (Skin and subcutaneous tissue disorders) | 28
rhinitis (Reproductive system and breast disorders) | 2
sinus tachycardia (Cardiac disorders) | 4
platelet count decreased (Investigations) | 4
thromboembolic event (Vascular disorders) | 3
upper respiratory infection (Infections and infestations) | 3
urinary frequency (Renal and urinary disorders) | 2
urinary tract infection (Infections and infestations) | 2
urticaria (Skin and subcutaneous tissue disorders) | 3
vomiting (Gastrointestinal disorders) | 11
weight loss (Investigations) | 5
vaccine site blisters (General disorders) | 5
vaccine site bruising (General disorders) | 3
vaccine site erythema (General disorders) | 31
vaccine site flares (General disorders) | 2
vaccine site induration (General disorders) | 37
vaccine site pruritus (General disorders) | 33
vaccine site tenderness (General disorders) | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigators (PIs) from participating sites must provide the Johns Hopkins PI with a copy of any proposed publication for review and comment at least 30 days prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT01896869/Prot_SAP_000.pdf